CLINICAL TRIAL: NCT00033098
Title: Cocaine-Metyrapone Interaction Study
Brief Title: Cocaine-Metyrapone Interaction Study - 1
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: Cincinnati VA Medical Center (U.S. Federal Agency)
Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-CTO-0006-1; NCT00024778 (obsolete NCT alias)
Record Dates: First submitted 2002-04-05; First posted 2002-04-08 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2003-08

CONDITIONS: Cocaine-Related Disorders; Infusions, Intravenous
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Metyrapone

INTERVENTIONS:
Drug: Metyrapone

SUMMARY:
The purpose of this study is to examine the safety of two consecutive days of metyrapone (MRP) in subjects who may use cocaine concurrently.

DETAILED DESCRIPTION:
To evaluate the safety of metyrapone (MRP) for using in an outpatient study in which participants would be given 2 750 mg doses of MRP per week. Secondary study goals are to evaluate the possible efficacy of MRP as a treatment for cocaine dependence and to compare 3 factors hypothesized to induce cocaine craving: cocaine cues, stress, and cocaine itself. This study will utilize a Double Blind, placebo-controlled crossover design with 3 factors: 1) medication 2) relapse trigger and 3) infusion for an 11 day in-patient treatment.

ELIGIBILITY:
Inclusion Criteria:

Male or Females between 18 and 45 yrs of age; cocaine dependence according to DSM-4; females of child-bearing potential must test non-pregnant and use adequate birth control; be able to provide consent, comply with protocol requirements and try to complete all study treatments.

Exclusion Criteria:

Additional criteria available during screening at the site.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12
Dates: Start 2001-11; Study Completion 2002-05

PRIMARY OUTCOMES:
Cocaine craving

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Winhusen, Ph.D., Principal Investigator — Cincinnati VA Medical Center
Locations (1):
- Cincinnati VA Medical Center, Cincinnati, Ohio, United States